CLINICAL TRIAL: NCT07165054
Title: Periodontal Pathogens and Atherom Plaque The Number of Mitochondrial DNA Copies
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ayşe Toraman, associate professor, Istanbul Saglik Bilimleri University
Other Study IDs: 1
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Inflammation; Biofilm; Endothelial Dysfunction; Oral Bacteria
MeSH Terms: interventions — Dental Plaque Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with endarterectomy
  Interventions: Other: atheroma plaque; Other: Dental plaque

INTERVENTIONS:
Other: atheroma plaque — Before the endarterectomy procedure, samples will be collected for study from some of the atheroma plaques routinely taken for pathology from patients.
Other: Dental plaque — Subgingival plaque samples will be collected from patients before the endarterectomy procedure.

SUMMARY:
Periodontitis is a chronic inflammatory disease of the tooth-supporting tissues characterized by the constant interaction of microorganisms in subgingival plaque and host defense mechanisms. Periodontitis is considered a focus of infection caused by oral bacteria, bacterial byproducts, or inflammatory mediators that can interact with other parts of the body via the bloodstream.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease of the tooth-supporting tissues characterized by the constant interaction of microorganisms in subgingival plaque and host defense mechanisms. Periodontitis is considered a focus of infection caused by oral bacteria, bacterial byproducts, or inflammatory mediators that can interact with other parts of the body via the bloodstream.

Periodontal bacteria produce endotoxins in the form of lipopolysaccharide (LPS). Circulating LPS reacts with Toll-like receptors, promoting the production of reactive oxygen species and phagocytosis in the intima layer. Oxidative stress has been reported to be associated with mtDNA copy number.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with endarterectomy
* Not receiving chemotherapy
* Not having received this treatment before

Exclusion Criteria:

* Having systemic infection
* Patients with severe heart disease

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endearterectomy diagnosed, dentate and edentulous patients
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Bacterial frequency (%) | Months 6-9 of the study
  The percentage of bacteria in the red complex in atheroma plaque and dental plaque is evaluated using polymerase chain reaction methods.

SECONDARY OUTCOMES:
Changes in mtDNA copy number (number) | Months 6-9 of the study
  Evaluation by means of quantitative polymerase chain reaction of mtDNA copy number in atheroma plaque
periodontal healths (mm) | 8 months
  Evaluation by means of periodontal indices such as PI, GI, BOP, PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Hamidiye Faculty of Dentistry, Department of Periodontology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No